CLINICAL TRIAL: NCT05889884
Title: Evaluation of the Dental Changes Associated With an Eight Units Extended Maxillary Fixed Retainer
Brief Title: Eight Units Extended Maxillary Fixed Retainer
Acronym: Extended FR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0479-8/2022
Record Dates: First submitted 2023-04-18; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2022-08

CONDITIONS: Orthodontic Retention
Keywords: Extended fixed retainer; 3D superimposition; Fixed retainers; PDL; Quality of life; Relapse
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Intervention Model Description: single arm prospect cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fixed retainer group (Experimental): test group who undergoes retention using extended maxillary fixed retainer
  Interventions: Device: Extended maxillary fixed retainer

INTERVENTIONS:
Device: Extended maxillary fixed retainer — Bonding extended maxillary fixed retainer from right first maxillary premolar to left maxillary first premolar for 6 months then assessment of relapse using 3D superimposition , little index , lateral cephalometric assessment along with PDL assessment with quality of life ,function and speech assessment

SUMMARY:
Assessment of dental changes associated with an eight-unit extended maxillary fixed retainer in 3D. monitoring PDL response and evaluation of patient's satisfaction ,quality of life and speech with extended maxillary fixed retainer

DETAILED DESCRIPTION:
single-arm prospective clinical trial will be conducted to assess of dental changes associated with an eight-unit extended maxillary fixed retainer in 3D. monitoring PDL response and evaluation of patient's satisfaction ,quality of life and speech with extended maxillary fixed retainer.

. Twenty-six patients who finished the active orthodontic treatment phase (14-28 years) will be recruited upon complying with the inclusion criteria. Eight-unit extended maxillary fixed retainer will be bonded to palatal surface of maxillary incisors, canines and first premolars, PDL assessment will be carried out and patient acceptance to the appliance through the valid questionnaire then the patients will be followed up for 6 months to document 3D post-treatment changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who finished the active orthodontic treatment and started the retention phase.
* Both genders.
* Extraction and non-extraction cases

Exclusion Criteria:

* Patients who had active transverse palatal expansion.
* Patients with active periodontal disease.
* Patients with systemic disease and bone diseases, or craniofacial syndromes, or the presence of cleft.
* Patients with abnormal surface or morphological tooth structure or restorations.

Ages: 14 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of dental changes | 6 months follow up
  3D Evaluation of the dental changes associated with an eight unit extended maxillary fixed retainer by superimposition of STL files before bonding and 6 months after bonding fixed retainer which is bonded directly after completion of active orthodontic phase, the changes in teeth position will be assessed by linear differences between the first stl and final stl file after superimposing them using medit software , on demand software ,creating linear measurement that calculate how teeth moved in antroposterior plane , transverse and vertical planes
lateral cephalometric changes assessment | 6months follow up
  evaluation of the changes of axial inclination of upper incisors before bonding fixed retainer and 6 months after bonding the retainer through measuring the axial inclination changes of upper incisors(u1-sn angle( upper 1 relation to cranial base ) , interincisal angle( angle between upper and lower incisors ) ,u1- FH angle( angle between upper incisor and Frankfort horizontal plane ) ,u1 to palatal plane angle (angle between upper incisor to palatal plane ), u1 to occlusal plane(angle between upper incisor and occlusal plane )

SECONDARY OUTCOMES:
PDL response through probing depth assessment | 6 months follow up
  Evaluation of PDL changes associated with the extended upper fixed retainer through comparison of probing depth changes before bonding the retainer and 6 months after bonding Probing depth:- is the distance from the gingival margin to the base of the sulcus or periodontal pocket. Normal range (1-3mm) the differences in probing depth readings will reflect either negative or no effect of fixed retainer on PDL
Gingival bleeding assessment | 6 months follow up
  Evaluation of PDL changes associated with the extended upper fixed retainer through calculating bleeding index before bonding and after 6 months of bonding fixed retainer Bleeding index:- method used to assess bleeding in the interdental tissues and gingiva.
  0: No bleeding. 1: Only one bleeding point appearing. 2: Several isolated bleeding points or a small blood area appearing. 3: Interdental triangle filled with blood soon after probing. 4: Profuse bleeding when probing, blood spreads towards the marginal gingiva.
  Changes in bleeding index will express effects of Fixed retainer on peridontium negatively or positively.
Plaque assessment | 6 months follow up
  Evaluation of PDL changes associated with the extended upper fixed retainer through calculating plaque index before bonding and after 6 months of bonding fixed retainer Plaque index:- method used to assess the amount of plaque on teeth.0 = No plaque in the gingival area. 1 = Separate flecks of plaque at the cervical margin of the tooth. 2 = A thin continuous band of plaque (up to 1 mm) at the cervical margin. 3 = Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.Changes in plaque index will express effects of Fixed retainer on PDL negatively or positively.
Gingival assessment | 6 months follow up
  Evaluation of PDL changes associated with the extended upper fixed retainer through calculating gingival index before bonding and after 6 months of bonding fixed retainer Gingival index:- method used to assess the severity of gingivitis.0 Normal gingiva Slight change in color, slight edema. No change on probing.1 Mild inflammation 2 Moderate inflammation Redness, edema, and glazing. Bleeding on probing. 3 Severe inflammation Marked redness and edema, ulceration. Tendency to spontaneous bleeding. Changes in gingival index readings will express effects of Fixed retainer on PDL negatively or positively.

OTHER OUTCOMES:
Quality of life assessment | 6 months follow up
  Evaluation of the quality of life ,through A-Oral Health Impact Profile (OHIP-14) valid and reliable tool for assessing oral health quality of life among the adults.The responses are rated on a 5-point Likert scale: 0-never,1-hardly ever,2-occasionally,3-fairly often,4-very often/every day. The OHIP-14 scores can range from 0 to 56 and are calculated by summing the ordinal values for the 14 items B-Acceptance questionnaire It consists of 10 incomplete statements,needed to be completed by patient's choice. The available answer choices were scored using a 6-point Likert scale. To help patients understand the answers, answers were accompanied by facial expression. Scores 5 to 0 were allocated to the answer choices from left to right.The higher scores the higher satisfaction with the item. The total score of this tool ranged from 0 to 55. A higher total score indicated that the problems of using the orthodontic appliance were better accepted by patient and motivation to continue.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed H abbas, BDS, Principal Investigator — Alexandria University; Essam M Abdallah, PHD, Study Director — Alexandria University; Nadia M Elharoni, PHD, Study Chair — Alexandria University; Eiman S marzouk, PHD, Study Chair — Alexandria University
Locations (1):
- Faculty of dentistry , Alexandria university, Alexandria, Egypt